CLINICAL TRIAL: NCT00188721
Title: Transillumination for Breast Cancer Risk Assessment
Brief Title: Breast Study to Learn More About the Application of Optical Transillumination Measurements to Assess Breast Cancer Risk and to Potentially Detect the Presence of Breast Cancer.
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Lothar Lilge, University Health Network
Other Study IDs: UHNREB#03-0462-CE; HC#96142
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Risk; Optical Transillumination Spectroscopy; Transillumination Breast Spectroscopy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Women with confirmed unilateral breast carcinoma or ductal carcinoma in situ (DCIS)
- 2: Women without radiological suspicious lesions, matched to cases by age (± 2.5 years), date of screening mammogram, and screening center.

SUMMARY:
This study aims to evaluate if a light based technique, called Transillumination Breast Spectroscopy (TIBS), can be used to construct a non-invasive breast cancer risk predictor which provides a better odds ratio than mammographic parenchymal density.

DETAILED DESCRIPTION:
In a previous cross sectional study in a group of women without breast cancer and with varying degrees of parenchymal density patterns, a strong association was demonstrated between Transillumination Breast Spectroscopy (TIBS) and x-ray derived mammographic density. From this, we expect that TIBS should also provide a comparable odds ratio (4-6) as mammographic density for breast cancer risk shown in other independent epidemiological studies. It is possible that TIBS may provide complementary information and a higher odds ratio if compared to the incidence of breast cancer. In contrast to mammography derived parenchymal density pattern, no historical TIBS data is available for a retrospective analysis and hence a cross sectional study within a group of screened women is proposed. We hypothesize that TIBS provides physical information about the breast tissue which can be used to construct a breast cancer risk predictor with an odd ratio > 6.

ELIGIBILITY:
Inclusion Criteria:

* Are in good health and capable of providing consent
* Are willing to come in to the Princess Margaret Hospital for a single visit to meet with a female research assistant

Exclusion Criteria:

* Have had breast augmentation or reduction
* Have a personal history of breast cancer
* Have had a previous bilateral fine needle aspiration or core biopsy
* Have a breast tattoo

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases and controls recruited from the Breast Imaging Clinic at Princess Margaret Hospital or the Marvelle Koffler Centre at Mount Sinai Hospital (Toronto, Ontario, Canada)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Lilge, PhD, Principal Investigator — Ontario Cancer Institute, University Health Network, Toronto, Ontario, Canada M5G 2M9; Department of Biophysics and Bioimaging, University of Toronto, Toronto, Ontario, Canada M5G 2M9
Locations (2):
- Canada (2):
  - Ontario Cancer Institute, Princess Maraget Hospital, Toronto, Ontario
  - Ontario Cancer Institute, Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Background] Blyschak K, Simick M, Jong R, Lilge L. Classification of breast tissue density by optical transillumination spectroscopy: optical and physiological effects governing predictive value. Med Phys. 2004 Jun;31(6):1398-414. doi: 10.1118/1.1738191. PMID 15259643
- [Background] Simick MK, Jong R, Wilson B, Lilge L. Non-ionizing near-infrared radiation transillumination spectroscopy for breast tissue density and assessment of breast cancer risk. J Biomed Opt. 2004 Jul-Aug;9(4):794-803. doi: 10.1117/1.1758269. PMID 15250768
- [Background] Blackmore KM, Knight JA, Jong R, Lilge L. Assessing breast tissue density by transillumination breast spectroscopy (TIBS): an intermediate indicator of cancer risk. Br J Radiol. 2007 Jul;80(955):545-56. doi: 10.1259/bjr/26858614. Epub 2007 May 30. PMID 17537757
- [Background] Simick MK, Lilge L. Optical transillumination spectroscopy to quantify parenchymal tissue density: an indicator for breast cancer risk. Br J Radiol. 2005 Nov;78(935):1009-17. doi: 10.1259/bjr/14696165. PMID 16249602